CLINICAL TRIAL: NCT00687765
Title: Phase I/II Study of the Poly (ADP-ribose) Polymerase-1 (PARP-1) Inhibitor BSI-201 in Patients With Newly Diagnosed Malignant Glioma
Brief Title: Study of the Poly (ADP-ribose) Polymerase-1 (PARP-1) Inhibitor BSI-201 in Patients With Newly Diagnosed Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11616; 20070104 (Other: BiPar); NCT00589576 (obsolete NCT alias)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2015-07

CONDITIONS: Glioblastoma
Keywords: patients with newly diagnosed glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — iniparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bsi-201 plus temozolomide

INTERVENTIONS:
Drug: bsi-201 plus temozolomide — BSI-201 given iv. 2x weekly, temozolomide given orally

SUMMARY:
The phase I portion of study is designed to determine the Maximum Tolerated Dose (MTD) of BSI-201 with two clinically relevant dosing regimens of temozolomide (TMZ). Secondary objectives in the phase I trial include determining the PK of BSI-201 in malignant glioma patients and correlating BSI-201 PK with degree of PARP-1 inhibition. A safety run-in will confirm the safety of BSI-201 added to standard TMZ and radiation therapy and the phase II portion of the study will assess the efficacy and tolerability of the MTD dose of BSI-201 with daily TMZ and radiation therapy followed by adjuvant TMZ in patients with newly diagnosed GBM and assess overall survival as the primary outcome measure. Information on each phase of the study will be listed when each phase opens for enrollment.

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age
2. Patients must have a Karnofsky performance status > 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
3. Patients must have the following hematologic, renal and liver function (i.e. Absolute neutrophil count > 1500/mm3, Platelets > 100,000/mm3, creatinine < 1.7 mg/dl, total bilirubin ≤ 1.5 mg/dl, transaminases < 4 times above the upper limits of the institutional normal
4. Patients must be able to provide written informed consent
5. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of childbearing potential must have a negative pregnancy test. The anti-proliferative activity of this experimental drug as well as the standard drug (temozolomide) may be harmful to the developing fetus or nursing infant
6. Patients must have a Mini Mental Status Exam score of > 15
7. Patients must have tumor tissue form completed and signed by a pathologist. See section 9.6 for details

Phase I Criteria (Phase I Patients ONLY)

1. Patients must have histologically proven supratentorial malignant glioma (anaplastic astrocytoma, anaplastic oligodendroglioma or glioblastoma multiforme)
2. Patients must have received at least 80% of planned temozolomide and radiation therapy with no grade 3 or grade 4 toxicity attributed to the temozolomide
3. Patients must have received planned treatment with radiation therapy and concomitant temozolomide at least 28 days but no more than 49 days prior to starting treatment on this study
4. Patients must have Gadolinium MRI or contrast CT scan within 28 days of starting treatment

Exclusion Criteria:

1. Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety
2. Patients who are pregnant or breast-feeding. The anti-proliferative activity of this experimental drug and temozolomide may be harmful to the developing fetus or nursing infant
3. Patients receiving concurrent therapy for their tumor (i.e. chemotherapeutics or investigational agents)
4. Patients with a concurrent or prior malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin. Patients who have been free of disease (any prior malignancy) for greater than five years are eligible for this study
5. Patients cannot be receiving cytochrome P450-inducing anticonvulsants (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital, primidone, oxcarbazepine) and must not have taken them for at least 10 days

Phase I Ineligibility Criteria (Phase I Patients ONLY)

1. Patients who have had repeat craniotomy for tumor therapy after receiving RT and TMZ treatment
2. Patients who received other chemotherapeutics or investigational agents in addition to their radiation therapy and concomitant temozolomide treatment. Patients who have received Gliadel wafers are eligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose (MTD) of BSI-201, administered as an IV infusion in patients with newly diagnosed malignant glioma when given with temozolomide (TMZ) after the completion of standard radiation therapy and concomitant TMZ | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- United States (8):
  - Research Site, Birmingham, Alabama
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Philadelphia, Pennsylvania